CLINICAL TRIAL: NCT02370771
Title: Proteomic Analysis in Sera From Patients With Erosive Hand Osteoarthritis
Acronym: PASEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/059/HP
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Erosive Hand Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patient with hand osteoarthritis (Experimental): Biological sampling and Radiographic evaluation of patient with erosive and non erosive hand osteoarthritis
  Interventions: Procedure: Biological sampling; Device: Radiographic evaluation

INTERVENTIONS:
Procedure: Biological sampling — Biological sampling to identify by label-free proteomic analysis of a combination of serum biomarkers in patients with Erosive and non erosive hand Osteoarthritis
Device: Radiographic evaluation — Radiographic assessments using Bone Mineral Analyser and Hand MRI will be done in patients with Erosive and non erosive hand Osteoarthritis

SUMMARY:
Hand osteoarthritis is a common phenotype of osteoarthritis which affects about 70 % of the elderly population. Usually considered as a minor illness, it nevertheless leads to an important functional impairment. The mechanism of this disease is still poorly known. Furthermore there are 2 different subtypes : erosive and non erosive hand osteoarthritis from which mechanisms may differ.

Methods:

This is a cross-sectional study recruiting patients with hand osteoarthritis addressed in consultation of rheumatology and plastic surgery in Rouen University Hospital.

Two groups of patients will be studied: 20 patients with non erosive subtype of hand osteoarthritis and 20 patients with erosive subtype of hand osteoarthritis.

A clinical evaluation of hand osteoarthritis will be performed. Blood sample for proteomic analysis will be taken. Hand MRI and Bone Mineral Analyser will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Less than 70 years old
* Diagnosis of hand osteoarthritis according to ACR criteria ACR after exclusion of thumb base osteoarthritis:

  1. Hand pain, aching or stiffness most of the days during the preceding month
  2. Hard tissue enlargement of at least two of 8 selected joints *
  3. Hard tissue enlargement of at least two distal interphalangeal joint
  4. Swelling of fewer than three metacarpophalangeal joint
  5. Deformity of at least one of 10 selected joints * Patients have to fulfil criteria 1, 2 AND 3 + 4 OR 5 * the 8 selected joints are the second and third distal interphalangeal joint and the second and third proximal interphalangeal of both hands Then confirm by experts' committee
* Exclusively symptomatic treatment
* For women of child-bearing age, use of an effective contraceptive method
* French spoken and read

Exclusion Criteria:

* Male gender
* More than 70 years old
* Hemochromatosis
* Inflammatory arthritis
* Cristal induced arthritis
* Active diseases such as infection or cancer
* Use of DMARDs
* Pregnant or breast-feeding woman

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06-09 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2019-11-17 (Actual)

PRIMARY OUTCOMES:
Quantification by label-free proteomic analysis of the serum of patients affected by hand osteoarthritis | day 1
  Assessments done using biological sampling

SECONDARY OUTCOMES:
Number of Erosion in patients affected by hand osteoarthritis | Day 1
  Number of Erosion in patients affected by hand osteoarthritis is evaluated using Bone Mineral Analyser

CONTACTS AND LOCATIONS:
Overall Officials: Gilles AVENEL, MD, Principal Investigator — UH Rouen
Locations (1):
- Rouen University Hospital, Rouen, France